CLINICAL TRIAL: NCT02483312
Title: Phase I Study of Autologous Acute Myelogenous Leukemia (AML) Cells Containing Lentivirus Engineering Expression of IL-12
Brief Title: A Study of (Interleukin-12) IL-12 in Patients With Acute Myelogenous Leukemia (AML)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ozmosis Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DDP-IL-12; OZM-068 (Other: Ozmosis Research Inc.)
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: Recurrent
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Interleukin-12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IL-12 (Experimental): A single dose of IL-12, given intravenously.
  Interventions: Biological: IL-12

INTERVENTIONS:
Biological: IL-12

SUMMARY:
This is a phase 1 study (the first stage in testing a new treatment to see how safe and tolerable the treatment is) which will include patients with acute myeloid leukemia (AML) that has either returned or has a more than a 70% chance of coming back and cannot have a bone marrow transplant.

This study will see whether modifying a patient's AML cells to produce IL-12 and giving it back to the patient is safe and useful in patients with AML that cannot have bone marrow transplants.

ELIGIBILITY:
Inclusion Criteria:

* Patient with AML and >=18 years of age.
* Agrees to participate in the study and signs the informed consent
* Viable cells are available for successful modification
* First or higher complete remission and have high risk features of relapse.
* Patients who have received prior treatment and are not in remission must have stable white blood cell count and are not receiving any chemotherapy or desiring further intensive treatment.
* Less than 10% blast cells in the bone marrow following induction or re-induction therapy and not desiring further intensive treatment.
* Acceptable creatinine, Aspartate transaminase (AST), Alkaline phosphatase (ALP), bilirubin lab results.
* Agree to use contraception
* Not pregnant
* Able to comply with study procedures

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status >2
* Known persistent infection
* Known central nervous system (CNS) disease
* Greater than 10% blasts in the bone marrow or circulating blast cells
* Life expectancy < 2 months
* Receiving any chemotherapy, corticosteroids, Cox2 inhibitors or any non-drug therapies with the intent of altering the immune response or kill leukemic cells within one week prior to infusion of IL-12, except azacytidine.
* Patients who are HIV positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2015-09; Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of side effects by type and severity | 2 years

SECONDARY OUTCOMES:
Levels of IL-12 | Day 28 to 2 years
  For patients who still show evidence of IL-12 producing AML cells on day 28, will be seen weekly for up to 2 years until there is no evidence of IL-12 producing cells
Levels of acute myeloid leukemia (AML) | Day 28 to 2 years
  For patients who still show evidence of IL-12 producing AML cells on day 28, will be seen weekly for up to 2 years until there is no evidence of IL-12 producing cells
Length of time patient is alive | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Sibai, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Centre Centre, Toronto, Ontario, Canada